CLINICAL TRIAL: NCT07178834
Title: Impact of a Tele-rehabilitation Program on People With Multiple Sclerosis: A Multicenter, Randomized, Single-blind Study.
Brief Title: Impact of a Tele-rehabilitation Program on People With Multiple Sclerosis
Acronym: Telerehab
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Multiple Sclerosis Center of Catalonia (Other)
Responsible Party: Principal Investigator, Edwin Roger Meza Murillo, DR, Multiple Sclerosis Center of Catalonia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR(AG)498/2024
Record Dates: First submitted 2025-07-04; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis
Keywords: Telerehabilitation; Rehabilitatiton; Patient-Reported Outcome Measures
MeSH Terms: conditions — Multiple Sclerosis | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: tele-rehabilitation (Experimental): This group will do online rehabilitation three times a week. Every two weeks, an assessment will be made to determine whether to increase the intensity of the exercise
  Interventions: Behavioral: Telerehab
- Control group: physical activity recommendations (No Intervention): This group will only have access to basic recommendations for physical activity.

INTERVENTIONS:
Behavioral: Telerehab — Adverse events are observed during online rehabilitation with computer vision technology in patients with MS.
  Other Names: Telerehabilitation; Intervention group
  Arms: Intervention group: tele-rehabilitation

SUMMARY:
The goal of this clinical trial is to assessing safety and the occurrence of adverse effects during tele-rehabilitation (TRHB) in people with multiple sclerosis with an EDSS score of 6.5 or lower. The main questions it aims to answer are:

* Intervention using TRHB is considered safe and without adverse effects.
* Intervention using TRHB has a high degree of self-adherence, an impact on physical activity levels and self-efficacy in exercise, and a positive effect on quality of life, mood, and perception of fatigue.

Researchers will compare the tele-rehabilitation with rehabilitation based solely on physical activity recommendations.

Participants will complete three weekly online rehabilitation sessions and must attend three follow-up visits.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) often entails a series of difficulties that cause some people to have high rates of absenteeism or even prevent them from benefiting from in-person rehabilitation treatments. The onset of the disease at a very young age, when the person is actively working or studying, the difficulty of balancing work and family life, mobility issues and lack of transportation, and geographical dispersion are some of the reasons why people with MS are not always able to access a neurorehabilitation center. Scientific evidence shows that functional and social barriers are the most common reasons why people do not adhere to rehabilitation. Home-based tele-rehabilitation (TRHB) is an alternative to rehabilitation in centers, allowing for remote supervision and the elimination of barriers. In addition, TRHB provides affected individuals and their families/caregivers with greater support in terms of care, mobility, and access to these services, and according to the World Health Organization (WHO), this type of assistance improves access to the healthcare system. There is a gap in research to identify the main adverse events related to tele-rehabilitation, and it is important to understand how adverse events, such as falls during physical therapy, are associated with the delivery of tele-rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with multiple sclerosis confirmed using the 2017 McDonald criteria.
* Patients who have the technological means to conduct online sessions and the autonomy to do so.
* Patients with cognitive capacity that allows them to sign the informed consent form.
* Patients with an internet connection and a device compatible with the Rehub tele-rehabilitation platform (desktop computer, laptop, or tablet).
* EDSS level less than or equal to 6.5.

Exclusion Criteria:

* Participants who are currently undergoing RHB at a center.
* Participants who have undergone RHB during the two months prior to the start of the program.
* Patients with physical or mental comorbidities that may limit their participation in the rehabilitation program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events | From enrollment to the end of treatment in week 8
  Adverse events such as falls, pain, fatigue, and others that may occur.

SECONDARY OUTCOMES:
Multiple Sclerosis Quality of Life 54 | (T1) baseline, (T2) after the 8 week, (T3) at 16 week.
  Quality of life scale (Min.0; Max.100). The higher the score, the better.
10 meters walking test | (T1) baseline, (T2) after the 8 week, (T3) at 16 week.
  The scale measures walking speed. There are no minimum or maximum measurements. The higher the reading, the better.
6 minute walking test | (T1) baseline, (T2) after the 8 week, (T3) at 16 week.
  The scale measures capacity for effort. There are no minimum or maximum measurements. The higher the score, the better.
Berg Balance Scale | (T1) baseline, (T2) after the 8 week, (T3) at 16 week.
  The scale measures the level of balance. Minimum measurement 0; maximum 56. The higher the reading, the better.

CONTACTS AND LOCATIONS:
Overall Officials: Edwin R Meza Murillo, Dr, Principal Investigator — Multiple Sclerosis Center of Catalonia
Locations (1):
- Multiple Sclerosis Center of Catalonia, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yau T, McIntyre M, Chan J, Bhogal D, Andreoli A, Bayley M, Leochico CFD, Kua A, Guo M, Munce S. Adverse events associated with the delivery of telerehabilitation: A scoping review protocol. PLoS One. 2024 Feb 21;19(2):e0297908. doi: 10.1371/journal.pone.0297908. eCollection 2024. PMID 38381732
- [Result] Doherty F, Lynch P, Powell P, Monaghan K. Feasibility and effectiveness of telerehabilitation on mobility and balance function in multiple sclerosis: A systematic review and meta-analysis. J Neurol Sci. 2024 Nov 15;466:123214. doi: 10.1016/j.jns.2024.123214. Epub 2024 Sep 4. PMID 39270413
- [Result] Xiang XM, Bernard J. Telehealth in Multiple Sclerosis Clinical Care and Research. Curr Neurol Neurosci Rep. 2021 Feb 28;21(4):14. doi: 10.1007/s11910-021-01103-4. PMID 33646409
- [Result] Harkey LC, Jung SM, Newton ER, Patterson A. Satisfacció del pacient amb la telesalud en entorns rurals: una revisió sistemàtica. Revista Internacional de Telerehabilitació. 2020;12(2):53-64. doi: 10.5195/ijt.2020.6303
- [Result] Fjeldstad-Pardo C, Thiessen A, Pardo G. Telerehabilitation in Multiple Sclerosis: Results of a Randomized Feasibility and Efficacy Pilot Study. Int J Telerehabil. 2018 Dec 11;10(2):55-64. doi: 10.5195/ijt.2018.6256. eCollection 2018 Fall. PMID 30588276

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-01-15): https://cdn.clinicaltrials.gov/large-docs/34/NCT07178834/Prot_SAP_000.pdf
  • Informed Consent Form (2025-01-15): https://cdn.clinicaltrials.gov/large-docs/34/NCT07178834/ICF_001.pdf